CLINICAL TRIAL: NCT06384326
Title: Comparison of Aesthetic Perception and Acceptability of Silver Diamine Fluoride Staining Between Spanish and Italian Parents.
Brief Title: Parental Perceptions and Acceptance of Silver Diamine Fluoride in Spain and Italy
Acronym: SDF
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Simone Bagattoni, Principal Investigator, University of Bologna
Other Study IDs: bagattoni3
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Comparative Study; Aesthetic Perception; Acceptability; SDF
Keywords: Silver Diamine Fluoride; Parental perceptions and acceptance; Comparative study; Spain and Italy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spanish parents: Spanish parents were recruited at the Department of Paediatric Dentistry of UIC between March 2023 and July 2023, accomplishing the second phase of the survey.
- Italian parents: Italian parents were recruited at the Unit of Dental Care for Special Needs Patients and Paediatric Dentistry at the University of Bologna, Bologna, Italy, and the Unit of Paediatric Dentistry at the University of Pisa, Pisa, Italy between September 2020 and March 2022

SUMMARY:
Assessing parental aesthetic acceptability of Silver Diamine Fluoride (SDF) staining is crucial for its potential implementation in paediatric dentistry. This study represents the third part of a wider project initially focused on evaluating SDF aesthetic acceptability in Italy, then comparing it between Spanish and Italian parents

DETAILED DESCRIPTION:
The aim of the present study was to compare aesthetic perceptions and acceptance of SDF pigmentation between Spanish and Italian parents, and assess weather acceptability is influenced by location, child's cooperation, or demographic background. A cross-sectional comparative study was conducted among 267 Spanish parents and 234 Italian parents whose children were attending three university dental clinics. A validated Italian version of the questionnaire "Parental perceptions of Silver Diamine Fluoride Dental Color Changes" was implemented. The questionnaire included sets of colored photographs showing both anterior and posterior teeth before and after SD treatment. Respondents were requested to provide their assessments based on the presented visual stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Spanish and Italian parents, for each group respectively
* Parents of healthy children or children with mild systemic disease. American Society of Anesthesiologists (ASA) status 1-2
* Parents of children under the age of 12 years
* Parents of children with previous caries experience in primary teeth
* Parents who consented to participate

Exclusion Criteria:

* No Spanish and Italian parents, for each group respectively
* Parents of children with ASA status ≥ 3
* Parents of children over the age of 12 years
* Parents of children without previous caries experience in primary teeth
* Parents who no consented to participate

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents awaiting their child's dental appointments at three distinct locations: for Italian parents the Unit of Dental Care for Special Needs Patients and Paediatric Dentistry at the University of Bologna, Bologna, Italy, and the Unit of Paediatric Dentistry at the University of Pisa, Pisa, Italy - for Spanish parents the Department of Paediatric Dentistry of the International University of Catalunya (UIC), Barcelona, Spain
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Comparison of SDF's overall acceptance between Spanish and Italian parents | Baseline
  Measurement tool: questionnaire. Specific questions focused on the general acceptability of the SDF staining for anterior and posterior teeth. Scores for levels of acceptability were 'unacceptable' (scoring 1), 'somewhat unacceptable' (scoring 2), 'somewhat acceptable' (scoring 3), and 'acceptable' (scoring 4). Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Comparison of SDF's specific acceptability in different scenarios of child's behavior between Spain and Italy | Baseline
  Measurement tool: questionnaire. Acceptance of SD treatment was evaluated by asking parents if they would allow the treatment to be done on their children in a context of hypothetical scenarios of child cooperation (child cooperative; child upset but could cooperate; child crying; child needs physical restraint; child screaming or kicking; child needs nitrous oxide sedation; child needs oral sedation; child needs general anesthesia). This assessment was carried out separately for anterior and posterior teeth. Scores for acceptance level were 'extremely unlikely' (scoring 1), 'somewhat unlikely' (scoring 2), 'somewhat likely' (scoring 3), and 'very likely' (scoring 4). Higher scores mean a better outcome.
Parental overall acceptability of SD staining according to demographic background | Baseline
  Measurement tool: questionnaire. Specific questions were strategically formulated to capture a comprehensive range of demographic variables of the participants, including factors such as age, education, and socioeconomic status. The findings from this analysis contribute valuable insights into the nuanced relationship between demographic characteristics and parental attitudes towards SD staining in Spain and Italy.

CONTACTS AND LOCATIONS:
Locations (1):
- Servizio di Assistenza Odontoiatrica per disabili in età evolutiva e di odontoiatria infantile, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cappiello MC, Duran AV, Crystal YO, Bagattoni S, Jimeno FG. Comparison of aesthetic perception and acceptability of silver diamine fluoride staining between Spanish and Italian parents. Sci Rep. 2025 Jan 27;15(1):3442. doi: 10.1038/s41598-025-87347-3. PMID 39870784